CLINICAL TRIAL: NCT03337698
Title: A Phase Ib/II, Open-Label, Multicenter, Randomized Umbrella Study Evaluating The Efficacy And Safety Of Multiple Immunotherapy-Based Treatment Combinations In Patients With Metastatic Non-Small Cell Lung Cancer (Morpheus-Lung)
Brief Title: A Study Of Multiple Immunotherapy-Based Treatment Combinations In Participants With Metastatic Non-Small Cell Lung Cancer (Morpheus- Non-Small Cell Lung Cancer)
Acronym: Morpheus Lung
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO39610; 2017-001267-21 (EudraCT Number)
Record Dates: First submitted 2017-11-07; First posted 2017-11-09 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — atezolizumab; cobimetinib; Docetaxel; ciforadenant; Pemetrexed; Carboplatin; Gemcitabine; Linagliptin; tocilizumab; ipatasertib; Bevacizumab; sacituzumab govitecan; Radiation; evolocumab; Tiragolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (23):
- Stage 1: Cohort 1: Atezolizumab (Active Comparator): Participants in the Atezolizumab arm will receive treatment (cycle length 21 days) until unacceptable toxicity or loss of clinical benefit.
  Participants who progressed on treatment, may have the option of receiving Atezolizumab + Pemetrexed + Carboplatin or Atezolizumab + Gemcitabine + Carboplatin treatment, provided they meet the eligibility criteria.
  Interventions: Drug: Atezolizumab
- Stage 1: Cohort 1: Atezolizumab + Cobimetinib (Experimental): Participants in the Atezolizumab + Cobimetinib arm will receive treatment (cycle length 28 days) until unacceptable toxicity or loss of clinical benefit.
  Participants who progressed on 1L treatment, may have the option of receiving Atezolizumab + Pemetrexed + Carboplatin or Atezolizumab + Gemcitabine + Carboplatin treatment, provided they meet the eligibility criteria.
  Participants who progressed on 2L/3L treatment, may have the option of receiving Atezolizumab + RO6958688, Atezolizumab + Docetaxel or Atezolizumab + Linagliptin treatment, provided they meet the eligibility criteria.
  Interventions: Drug: Atezolizumab; Drug: Cobimetinib
- Stage 1: Cohort 1: Atezolizumab + RO6958688 (Experimental): Participants in the Atezolizumab + RO6958688 arm will receive treatment (cycle length 21 days) until unacceptable toxicity or loss of clinical benefit.
  Participants who progressed on 1L treatment, may have the option of receiving Atezolizumab + Pemetrexed + Carboplatin or Atezolizumab + Gemcitabine + Carboplatin treatment, provided they meet the eligibility criteria.
  Participants who progressed on 2L/3L treatment, may have the option of receiving Atezolizumab + Docetaxel treatment or Atezolizumab + Linagliptin treatment, provided they meet the eligibility criteria.
  Interventions: Drug: Atezolizumab; Drug: RO6958688; Drug: Tocilizumab
- Stage 1: Cohort 2: Docetaxel (Active Comparator): Participants in the Docetaxel arm will receive treatment (cycle length 21 days) until unacceptable toxicity or disease progression.
  Participants who progressed on treatment may have the option of receiving Atezolizumab + RO6958688 or Atezolizumab + Linagliptin treatment, provided they meet the eligibility criteria.
  Interventions: Drug: Docetaxel
- Stage 1: Cohort 2: Atezolizumab + Cobimetinib (Experimental): Participants in the Atezolizumab + Cobimetinib arm will receive treatment (cycle length 28 days) until unacceptable toxicity or loss of clinical benefit.
  Participants who progressed on treatment, may have the option of receiving Atezolizumab + Pemetrexed + Carboplatin, Atezolizumab + Gemcitabine + Carboplatin, Atezolizumab + RO6958688, Atezolizumab + Docetaxel or Atezolizumab + Linagliptin treatment, provided they meet the eligibility criteria.
  Interventions: Drug: Atezolizumab; Drug: Cobimetinib
- Stage 1: Cohort 2: Atezolizumab + CPI-444 (Experimental): Participants in the Atezolizumab + CPI-444 arm will receive treatment (cycle length 21 days) until unacceptable toxicity or loss of clinical benefit.
  Participants who progressed on treatment, may have the option of receiving Atezolizumab + RO6958688, Atezolizumab + Docetaxel or Atezolizumab + Linagliptin treatment, provided they meet the eligibility criteria.
  Interventions: Drug: Atezolizumab; Drug: CPI-444
- Stage 1: Cohort 2: Atezolizumab + RO6958688 (Experimental): Participants in the Atezolizumab + RO6958688 arm will receive treatment (cycle length 21 days) until unacceptable toxicity or loss of clinical benefit.
  Participants who progressed on treatment, may have the option of receiving Atezolizumab + Pemetrexed + Carboplatin, Atezolizumab + Gemcitabine + Carboplatin, Atezolizumab + Docetaxel or Atezolizumab + Linagliptin treatment, provided they meet the eligibility criteria.
  Interventions: Drug: Atezolizumab; Drug: RO6958688; Drug: Tocilizumab
- Stage 1: Cohort 2: Atezolizumab + Ipatasertib (Experimental): Participants in the Atezolizumab + Ipatasertib arm will receive treatment (cycle length 28 days) until unacceptable toxicity or loss of clinical benefit.
  Participants who progressed on treatment, may have the option of receiving Atezolizumab + Docetaxel treatment or Atezolizumab + Linagliptin treatment, provided they meet the eligibility criteria.
  Interventions: Drug: Atezolizumab; Drug: Ipatasertib
- Stage 1: Cohort 2: Atezolizumab + Docetaxel (Experimental): Participants in Atezolizumab + Docetaxel arm will receive treatment (cycle length 21 days) until unacceptable toxicity or loss of clinical benefit.
  Participants who progressed on treatment, may have the option of receiving Atezolizumab + Linagliptin treatment, provided they meet the eligibility criteria.
  Interventions: Drug: Atezolizumab; Drug: Docetaxel
- Stage 1: Cohort 2: Atezolizumab + Bevacizumab (Experimental): Participants in Atezolizumab + Bevacizumab arm will receive treatment (cycle length 21 days) until unacceptable toxicity or loss of clinical benefit.
  Participants who progressed on treatment, may have the option of receiving Atezolizumab + Docetaxel or Atezolizumab + Linagliptin treatment, provided they meet the eligibility criteria.
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab
- Stage 2: Cohort 1: Atezolizumab + Pemetrexed + Carboplatin (Experimental): Participants in the Atezolizumab + Pemetrexed + Carboplatin arm will receive treatment (cycle length 21 days) until unacceptable toxicity or loss of clinical benefit.
  Interventions: Drug: Atezolizumab; Drug: Pemetrexed; Drug: Carboplatin
- Stage 2: Cohort 1: Atezolizumab + Gemcitabine + Carboplatin (Experimental): Participants in the Atezolizumab + Gemcitabine + Carboplatin arm will receive treatment (cycle length 21 days) until unacceptable toxicity or loss of clinical benefit.
  Interventions: Drug: Atezolizumab; Drug: Carboplatin; Drug: Gemcitabine
- Stage 2: Cohort 2: Atezolizumab + RO6958688 (Experimental): Participants in the Atezolizumab + RO6958688 arm will receive treatment (cycle length 21 days) until unacceptable toxicity or loss of clinical benefit.
  Interventions: Drug: Atezolizumab; Drug: RO6958688; Drug: Tocilizumab
- Stage 2: Cohort 2: Atezolizumab + Docetaxel (Experimental): Participants in the Atezolizumab + Docetaxel arm will receive treatment (cycle length 21 days) until unacceptable toxicity or loss of clinical benefit.
  Participants who have received treatment with Atezolizumab + Docetaxel in Stage 1 will not receive this treatment in Stage 2.
  Interventions: Drug: Atezolizumab; Drug: Docetaxel
- Stage 2: Cohort 2: Atezolizumab + Linagliptin (Experimental): Participants in the Atezolizumab + Linagliptin arm will receive treatment (cycle length 21 days) until unacceptable toxicity or loss of clinical benefit.
  Interventions: Drug: Atezolizumab; Drug: Linagliptin
- Stage 1: Cohort 2: Atezolizumab + Sacituzumab Govitecan (Experimental): Participants in the Atezolizumab + Sacituzumab Govitecan arm will receive treatment (cycle length 21 days) until unacceptable toxicity or loss of clinical benefit.
  Interventions: Drug: Atezolizumab; Drug: Sacituzumab Govitecan
- Stage 1: Cohort 2: Atezolizumab + Bevacizumab + Radiotherapy (Experimental): Participants in the Atezolizumab + Bevacizumab + Radioatherapy arm will receive treatment (cycle length 21 days) until unacceptable toxicity or loss of clinical benefit.
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab; Other: Radiation
- Stage 1: Cohort 2: Atezolizumab + Evolocumab (Experimental): Participants in the Atezolizumab + Evolocumab arm will receive treatment (cycle length 28 days) until unacceptable toxicity or loss of clinical benefit.
  Interventions: Drug: Atezolizumab; Drug: Evolocumab
- Stage 1: Cohort 1: Atezolizumab + Tiragolumab (Active Comparator): Participants in the Atezolizumab + Tiragolumab arm will receive treatment (cycle length 21 days) until unacceptable toxicity or loss of clinical benefit.
  Interventions: Drug: Atezolizumab; Drug: Tiragolumab
- Stage 1: Cohort 1: Atezolizumab + Tiragolumab + XL092 (Zanzalintinib) (Experimental): Participants in the Atezolizumab + Tiragolumab + XL092 arm will receive treatment (cycle length 21 days) until unacceptable toxicity or loss of clinical benefit.
  Interventions: Drug: Atezolizumab; Drug: Tiragolumab; Drug: XL092
- Stage 1: Cohort 2: Atezolizumab + Camonsertib (Experimental): Participants in the Atezolizumab + Camonsertib arm will receive treatment (cycle length 21 days) until unacceptable toxicity or loss of clinical benefit.
  Interventions: Drug: Atezolizumab; Drug: Camonsertib
- Stage 1: Cohort 2: Atezolizumab + Bevacizumab + Camonsertib (Experimental): Participants in the Atezolizumab + Bevacizumab + Comonsertib arm will receive treatment (cycle length 21 days) until unacceptable toxicity or loss of clinical benefit.
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab; Drug: Camonsertib
- Stage 1: Cohort 2: Atezolizumab + Bevacizumab + Tiragolumab (Experimental): Participants in the Atezolizumab + Bevacizumab + Tiragolumab arm will receive treatment (cycle length 21 days) until unacceptable toxicity or loss of clinical benefit.
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab; Drug: Tiragolumab

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab is administered by IV on Day 1 of each 21 day cycle or on Days 1 and 15 of each 28 day cycle.
  Arms: Stage 1: Cohort 1: Atezolizumab; Stage 1: Cohort 1: Atezolizumab + Cobimetinib; Stage 1: Cohort 1: Atezolizumab + RO6958688; Stage 1: Cohort 1: Atezolizumab + Tiragolumab; Stage 1: Cohort 1: Atezolizumab + Tiragolumab + XL092 (Zanzalintinib); Stage 1: Cohort 2: Atezolizumab + Bevacizumab; Stage 1: Cohort 2: Atezolizumab + Bevacizumab + Camonsertib; Stage 1: Cohort 2: Atezolizumab + Bevacizumab + Radiotherapy; Stage 1: Cohort 2: Atezolizumab + Bevacizumab + Tiragolumab; Stage 1: Cohort 2: Atezolizumab + CPI-444; Stage 1: Cohort 2: Atezolizumab + Camonsertib; Stage 1: Cohort 2: Atezolizumab + Cobimetinib; Stage 1: Cohort 2: Atezolizumab + Docetaxel; Stage 1: Cohort 2: Atezolizumab + Evolocumab; Stage 1: Cohort 2: Atezolizumab + Ipatasertib; Stage 1: Cohort 2: Atezolizumab + RO6958688; Stage 1: Cohort 2: Atezolizumab + Sacituzumab Govitecan; Stage 2: Cohort 1: Atezolizumab + Gemcitabine + Carboplatin; Stage 2: Cohort 1: Atezolizumab + Pemetrexed + Carboplatin; Stage 2: Cohort 2: Atezolizumab + Docetaxel; Stage 2: Cohort 2: Atezolizumab + Linagliptin; Stage 2: Cohort 2: Atezolizumab + RO6958688
Drug: Cobimetinib — Cobimetinib is administered orally on Days 1-21 of a 28 day cycle.
  Arms: Stage 1: Cohort 1: Atezolizumab + Cobimetinib; Stage 1: Cohort 2: Atezolizumab + Cobimetinib
Drug: RO6958688 — Cycle 1:
  RO6958688 is administered by IV infusion on Days 1, 8, and 15 of a 21 day cycle at increasing dosage.
  Subsequent cycles:
  RO6958688 is administered by IV infusion on Days 1, 8, and 15 of a 21 day cycle.
  Arms: Stage 1: Cohort 1: Atezolizumab + RO6958688; Stage 1: Cohort 2: Atezolizumab + RO6958688; Stage 2: Cohort 2: Atezolizumab + RO6958688
Drug: Docetaxel — Docetaxel is administered by IV on Day 1 of each 21 day cycle.
  Arms: Stage 1: Cohort 2: Atezolizumab + Docetaxel; Stage 1: Cohort 2: Docetaxel; Stage 2: Cohort 2: Atezolizumab + Docetaxel
Drug: CPI-444 — CPI-444 is administered orally twice daily on Days 1- 21, of a 21 day cycle.
  Arms: Stage 1: Cohort 2: Atezolizumab + CPI-444
Drug: Pemetrexed — Pemetrexed is administered by IV on Day 1 of a 21 day cycle.
  Arms: Stage 2: Cohort 1: Atezolizumab + Pemetrexed + Carboplatin
Drug: Carboplatin — Carboplatin is administered by IV on day 1 of the first 4 or 6 cycles out of a 21 day cycle.
  Arms: Stage 2: Cohort 1: Atezolizumab + Gemcitabine + Carboplatin; Stage 2: Cohort 1: Atezolizumab + Pemetrexed + Carboplatin
Drug: Gemcitabine — Gemcitabine is administered by IV on Days 1 and 8 of the first 4 or 6 cycles out of a 21 day cycle.
  Arms: Stage 2: Cohort 1: Atezolizumab + Gemcitabine + Carboplatin
Drug: Linagliptin — Linagliptin is administered orally once daily on Days 1 to 21 out of a 21 day cycle.
  Arms: Stage 2: Cohort 2: Atezolizumab + Linagliptin
Drug: Tocilizumab — Tocilizumab is administered for the management of cytokine-release syndrome in the RO6958688-containing arms.
  Arms: Stage 1: Cohort 1: Atezolizumab + RO6958688; Stage 1: Cohort 2: Atezolizumab + RO6958688; Stage 2: Cohort 2: Atezolizumab + RO6958688
Drug: Ipatasertib — Ipatasertib will be administered orally once a day on Days 1-21 of each 28-day cycle.
  Arms: Stage 1: Cohort 2: Atezolizumab + Ipatasertib
Drug: Bevacizumab — Bevacizumab is administered by IV on Day 1 of each 21-day cycle.
  Arms: Stage 1: Cohort 2: Atezolizumab + Bevacizumab; Stage 1: Cohort 2: Atezolizumab + Bevacizumab + Camonsertib; Stage 1: Cohort 2: Atezolizumab + Bevacizumab + Radiotherapy; Stage 1: Cohort 2: Atezolizumab + Bevacizumab + Tiragolumab
Drug: Sacituzumab Govitecan — Sacituzumab Govitecan is administered by IV on Day 1 and 8 of each 21-day cycle.
  Arms: Stage 1: Cohort 2: Atezolizumab + Sacituzumab Govitecan
Other: Radiation — Radiotherapy up to 21 days
  Arms: Stage 1: Cohort 2: Atezolizumab + Bevacizumab + Radiotherapy
Drug: Evolocumab — Evolocumab is administered subcutaneously at a dose of 140 mg on Days 1 and 15 of each 28-day cycle.
  Arms: Stage 1: Cohort 2: Atezolizumab + Evolocumab
Drug: Tiragolumab — Tiragolumab is administered on Day 1 of each 21 day cycle.
  Arms: Stage 1: Cohort 1: Atezolizumab + Tiragolumab; Stage 1: Cohort 1: Atezolizumab + Tiragolumab + XL092 (Zanzalintinib); Stage 1: Cohort 2: Atezolizumab + Bevacizumab + Tiragolumab
Drug: XL092 — XL092 is administered orally once a day on Day 1 to Day 21 of a 21 day cycle.
  Other Names: Zanzalintinib
  Arms: Stage 1: Cohort 1: Atezolizumab + Tiragolumab + XL092 (Zanzalintinib)
Drug: Camonsertib — Camonsertib is administered orally on Days 1-3, Days 8-10 of a 21 day cycle.
  Arms: Stage 1: Cohort 2: Atezolizumab + Bevacizumab + Camonsertib; Stage 1: Cohort 2: Atezolizumab + Camonsertib

SUMMARY:
This study will evaluate the efficacy, safety, and pharmacokinetics of immunotherapy-based treatment combinations in participants with metastatic non-small cell lung cancer (NSCLC).

Two cohorts will be enrolled in parallel in this study: Cohort 1 will consist of participants with tumor PD-L1 expression who have received no prior systemic therapy for metastatic NSCLC, and Cohort 2 will consist of participants who experienced disease progression during or following treatment with a platinum-containing regimen and a PD-L1/PD-1 checkpoint inhibitor, given in combination as one line of therapy or as two separate lines of therapy, regardless of PD-L1 expression. In each cohort, eligible participants will initially be assigned to one of several treatment arms (Stage 1). Participants who experience disease progression, loss of clinical benefit, or unacceptable toxicity during Stage 1 may be eligible to continue treatment with a different treatment regimen (Stage 2).

ELIGIBILITY:
General Inclusion Criteria

* Eastern Cooperative Oncology Group (ECOG) performance Status of 0 or 1
* Life expectancy greater than or equal to 3 months
* Histologically or cytologically confirmed metastatic, non-squamous or squamous Non-Small Cell Lung Cancer (NSCLC)
* Measurable disease (at least one target lesion)
* Adequate hematologic and end-organ function
* Tumor accessible for biopsy
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures and agreement to refrain from donating eggs as outlined for each specific treatment arm
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm, as outlined for each specific treatment arm

Inclusion Criteria for Cohort 1

* No prior systemic therapy for metastatic NSCLC
* High tumor PD-L1 expression, defined as Tumor Proportion Score (TPS) or TCs >= 50% or TC3

Inclusion Criteria for Cohort 2

- Disease progression during or following treatment for metastatic or locally advanced, inoperable NSCLC

Exclusion Criteria

* Prior allogeneic stem cell or solid organ transplantation
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently)
* Symptomatic, untreated, or actively progressing central nervous system (CNS) metastases
* History of leptomeningeal disease
* Active or history of autoimmune disease or immune deficiency
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography scan
* History of malignancy other than NSCLC within 2 years prior to screening
* Active tuberculosis
* Severe infection within 4 weeks prior to initiation of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2017-12-27 (Actual); Primary Completion 2025-10-14 (Actual); Study Completion 2025-11-25 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Objective Response | Every 6 weeks (starting on Day 1, Cycle 1) for the first 48 weeks and then every 6 or 12 weeks thereafter

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | Randomization to the first occurrence of disease progression or death from any cause (up to approximately 8 years)
Overall Survival After Randomization | Randomization to death from any cause (up to approximately 8 years)
Percentage of Participants Who Are Alive at Month 6 and at Month 12 | Month 6, Month 12
Duration of Response | First occurrence of a documented objective response to disease progression or death (up to approximately 8 years)
Disease Control | Randomization to the first occurrence of disease progression or death from any cause (up to approximately 8 years)
Percentage of Participants with Adverse Events | Baseline through the end of the study (approximately 8 years)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (29):
- United States (4):
  - Comprehensive Cancer Centers of Nevada (CCCN) - Central Valley, Las Vegas, Nevada
  - Columbia University Medical Center, New York, New York
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - SCRI Oncology Partners, Nashville, Tennessee
- Australia (2):
  - Blacktown Hospital, Blacktown, New South Wales
  - Peter Mac Callum Cancer Center, East Melbourne, Victoria
- France (6):
  - Centre Georges Francois Leclerc, Dijon
  - Centre Léon Bérard, Lyon
  - Hopital de la Timone, Marseille
  - Institut Régional du Cancer de Montpellier, Montpellier
  - Institut De Cancerologie De L'Ouest, Saint-Herblain
  - Institut Universitaire du Cancer de Toulouse-Oncopole, Toulouse
- Israel (3):
  - Rambam Medical Center, Haifa
  - Rabin Medical Center, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
- South Korea (4):
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Korea University Guro Hospital, Seoul
  - University of Ulsan College of Medicine - Asan Medical Center (AMC) - Asan Cancer Center (ACC), Songpa-gu
- Spain (7):
  - Clínica Universidad de Navarra, Pamplona, Navarre
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Fundación Jimenez Díaz, Madrid
  - Hospital Universitario HM Sanchinarro-CIOCC, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital Clinico Universitario de Valencia, Valencia
- United Kingdom (3):
  - Barts Cancer Institute, London
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne
  - Royal Marsden Hospital, Sutton

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing